CLINICAL TRIAL: NCT06076460
Title: Early Total Enteral Feeding Versus Convention Enteral Feeding in Preterm Neonates Between 27 to 32 Weeks of Gestation: A Randomized Control Trial
Brief Title: Early Total Enteral Feeding Versus Convention Enteral Feeding in Preterm Infants 27-32 Weeks of Gestation
Acronym: ETEFVsCEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Sushma Nangia, M.D., Dr Sushma Nangia, Director Professor & Head, Neonatology, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: LHMC/IEC/2021/03/68
Record Dates: First submitted 2023-08-31; First posted 2023-10-10 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Very Preterm Maturity of Infant; Enteral Feeding Intolerance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Total Enteral Feeding (Experimental): Mom's milk or donor milk at 80 ml/kg/day after randomization within the first 2 hours
  Interventions: Other: Early Total Enteral Feeding
- Conventional Enteral Feeding (Active Comparator): Mom's milk or donor milk at 20 ml/kg/day and rest of the requirement as Total parenteral nutrition after randomization within the first 2 hours.
  Interventions: Other: Conventional Enteral Feeding

INTERVENTIONS:
Other: Early Total Enteral Feeding — This group will receive enteral feeding volumes at a rate of 80 ml/kg/day starting within the first two hours after birth. Volumes will increased by 20 ml/kg/day till day 4 (total 140 ml/kg/d) and then 150ml/kg/day on day 5.
  Arms: Early Total Enteral Feeding
Other: Conventional Enteral Feeding — This group will receive enteral feeding volumes at a rate of 20 ml/kg/day starting within the first two hours after birth and rest of the daily requirement as Total parenteral nutrition. Volumes will be increased by 20 ml/kg/day till day 3 and thereafter by 30 ml/kg/d till 150ml/kg/day on day 6.
  Arms: Conventional Enteral Feeding

SUMMARY:
The objective of the study is to compare the time of attainment of full enteral feeds in preterm neonates between 27-32 weeks of gestation started on early total enteral feeding (ETEF) with those started on conventional enteral feeding (CEF).

DETAILED DESCRIPTION:
Enrolled participants will be randomly assigned to one of two study groups: 1) early total enteral feeding (ETEF) or 2) conventional enteral feeding (CEF). Regardless of study group assignment, mother's own breast milk (MOM) is the feed of choice and donor human milk is being offered if the MOM is not enough to complete the intervention as assigned

Intervention group: Feeds will be initiated with a target volume of 80 ml/kg/day starting within the first two hours after birth. Volumes will increased by 20 ml/kg/day till day 4 (total 140 ml/kg/d) and then 150ml/kg/day on day 5.

Control group: This group will receive enteral feeding volumes at a rate of 20 ml/kg/day starting within the first two hours after birth and rest of the daily requirement as Total parenteral nutrition. Volumes will be increased by 20 ml/kg/day till day 3 and thereafter by 30 ml/kg/d till 150ml/kg/day on day 6.

ELIGIBILITY:
Inclusion Criteria:

Preterm neonate with gestational age of 27-32 weeks

Exclusion Criteria:

1. Antenatally diagnosed GI malformation
2. Baby born with absence or reversal of end diastolic flow on antenatal umbilical artery Doppler.
3. Presence of major congenital anomalies at birth
4. Need of vasopressor support at the time of randomization
5. Requiring Positive Pressure Ventilation > 60 sec with APGAR score < 4 at 1 minute

Max Age: 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 183 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-10 (Actual)

PRIMARY OUTCOMES:
Time of attainment of full enteral feeds (150ml/kg/day) during the first 28 days after birth | Birth to 28 days
  Days to attain full feeds during the first 28 days after birth

SECONDARY OUTCOMES:
Number of episodes of feeding intolerance | From Randomization till 28 days after birth
  Feed intolerance will be defined as any one or more of the following a) Vomiting 3 or more in any 24 hour period, b) Any episode of blood stained or bilious vomiting, c) Abdominal girth(AG) increase >2 cm (with pre-feed aspirate >25%), abdominal wall erythema or tenderness, gross or occult blood in stools
Incidence of Necrotising Enterocolitis | From Randomization till 28 days after birth
  Diagnosis of necrotizing enterocolitis any stage
Incidence of Sepsis | From randomization till 28 days after birth
  Sepsis will be defined as any one of the following in a symptomatic neonate a) Culture positive sepsis b) Sepsis screen positive, c) Strong clinical suspicion such as sclerema, shock or clinical deterioration on supportive therapy which warrants initiation of antibiotics (clinician decision)
Total duration of intravenous fluid usage | From randomization till 28 days after birth
  Duration in completed days for which infant required parenteral fluid support
Time of regaining birth weight | From randomization till 28 days after birth
  Duration in completed days required to regain birth weight
Total duration of hospital stay | From randomization till 2 months after birth
  Duration in completed days required for treatment till discharge home or till death
Weight gain per kg per day at 1 month of age | Birth to 30 days
  The weight in grams at one month of age minus the birth weight divided by the average weight (average weight =birth weight +Weight at 1 month age divided by 2) further divided by 30
Extrauterine growth retardation (EUGR) | Till 36 weeks Postmenstrual age
  Weight of the infants at 36 weeks Postmenstrual age or at discharge (if earlier) below the 10th centile for age

CONTACTS AND LOCATIONS:
Overall Officials: Sushma Nangia, DM (NEO), Study Chair — Lady Hardinge Medical College
Locations (1):
- Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walsh V, Brown JVE, Copperthwaite BR, Oddie SJ, McGuire W. Early full enteral feeding for preterm or low birth weight infants. Cochrane Database Syst Rev. 2020 Dec 27;12(12):CD013542. doi: 10.1002/14651858.CD013542.pub2. PMID 33368149
- [Background] Nangia S, Bishnoi A, Goel A, Mandal P, Tiwari S, Saili A. Early Total Enteral Feeding in Stable Very Low Birth Weight Infants: A Before and After Study. J Trop Pediatr. 2018 Feb 1;64(1):24-30. doi: 10.1093/tropej/fmx023. PMID 28431170